CLINICAL TRIAL: NCT06750445
Title: The Safety and Efficacy of Fluoxetine for Treatment of Refractory Constipation
Brief Title: Fluoxetine for Refractory Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhifeng Zhao, PhD (Other)
Responsible Party: Sponsor-Investigator, Zhifeng Zhao, PhD, Dr., Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJLL-KY20222069
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-12

CONDITIONS: Refractory Constipation
MeSH Terms: conditions — Constipation | interventions — Fluoxetine; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoxetine Treatment Group (Experimental): Patients in the fluoxetine group received oral fluoxetine starting at 40 mg/day for six months. The dose could be increased to 60 mg/day if symptoms persisted or reduced if mild adverse effects (e.g., dizziness, nausea, tremors) occurred. Treatment was discontinued if serious adverse reactions developed or if no improvement was observed after dose escalation. Compliance and treatment progress were monitored via telephone follow-ups. For patients unable to have a bowel movement for three consecutive days or experiencing intolerable symptoms, polyethylene glycol (PEG, 10 g) was provided as rescue medication. Bowel movements within 24 hours of rescue medication use were excluded from the count of complete spontaneous bowel movements (CSBM).
  Interventions: Drug: Fluoxetine
- PEG Treatment Group (Active Comparator): The control group (PEG) used polyethylene glycol as a rescue medication under the same conditions, following similar monitoring and follow-up procedures.
  Interventions: Drug: Polyethylene Glycol 400 0.4%

INTERVENTIONS:
Drug: Fluoxetine — Patients in the fluoxetine group received oral fluoxetine starting at 40 mg/day for six months. Treatment was discontinued if serious adverse reactions developed or if no improvement was observed after dose escalation. Compliance and treatment progress were monitored via telephone follow-ups. For patients unable to have a bowel movement for three consecutive days or experiencing intolerable symptoms, polyethylene glycol (PEG, 10 g) was provided as rescue medication. Bowel movements within 24 hours of rescue medication use were excluded from the count of complete spontaneous bowel movements (CSBM).
  Other Names: polyethylene glycol
  Arms: Fluoxetine Treatment Group
Drug: Polyethylene Glycol 400 0.4% — The control group (PEG) used polyethylene glycol as a rescue medication under the same conditions, following similar monitoring and follow-up procedures.
  Arms: PEG Treatment Group

SUMMARY:
The goal of this clinical trial is to learn if fluoxetine works to treat refractory constipation . It will also learn about the safety of fluoxetine. The main questions it aims to answer are:

Does fluoxetine increase the number of completely spontaneous bowel movements (CSBMs) per week? What medical problems do participants have when taking fluoxetine? Does fluoxetine improve psychological symptoms such as anxiety and depression in participants with refractory constipation? Researchers will compare fluoxetine to polyethylene glycol (PEG, a commonly used laxative) to see if fluoxetine works to treat refractory constipation.

Participants will:

Take fluoxetine (40 mg/day) or polyethylene glycol (once daily) for 6 months. Visit the clinic at baseline, and at 1 month, 3 months, and 6 months for checkups and tests.

Record their bowel movements and any changes in symptoms, including anxiety, depression, and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. individuals aged 18 to 70 years;
2. patients meeting the Rome IV diagnostic criteria for chronic constipation, defined by at least two symptoms: straining, lumpy or hard stools (Bristol Stool Scale types 1-2), incomplete evacuation, anorectal obstruction, need for manual maneuvers, or spontaneous bowel movements occurring less than three times per week. These symptoms must have persisted for a minimum of six months, with the diagnostic criteria being met for at least the past three months;
3. refractory constipation, defined as the use of at least three medications (including osmotic agents, laxatives, prokinetics, biofeedback and probiotics, surgery) for more than three months, with unsatisfactory treatment outcomes;
4. patients present indications for fluoxetine, such as comorbid depression;
5. patients who voluntarily provided informed consent prior to enrollment.

Exclusion Criteria:

1. women who are pregnant or lactating;
2. presence of cardiovascular conditions, organ dysfunction, immune disorders, or infections;
3. concurrent gastrointestinal organic conditions such as tuberculosis, polyps, Crohn's disease, tumors, etc.;
4. prior abdominal surgeries;
5. use of psychotropic medications; 6) diagnosis of hypothyroidism or Parkinson's disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a CSBM of 3 or more per week | baseline, six months after treatment
  The primary endpoint of this study is the proportion of patients achieving a weekly frequency of three or more complete spontaneous bowel movements (CSBMs) after six months of treatment. A CSBM is defined as a bowel movement that occurs without the use of rescue medication (e.g., polyethylene glycol) within the preceding 24 hours. This endpoint aims to evaluate the efficacy of fluoxetine in improving bowel function in patients with refractory constipation as compared to the control group.

SECONDARY OUTCOMES:
Mean number of spontaneous bowel movements (SBMs) per week | baseline, 1 month, 3 months, 6 months
Mean number of complete spontaneous bowel movements (CSBMs) per week | baseline, 1 month, 3 months, 6 months
Stool consistency (Bristol Stool Form Scale, BSFS, scores of 3-5) | baseline, 1 month, 3 months, 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - The First Affiliated Hospital of the Fourth Military Medical University, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No